CLINICAL TRIAL: NCT01674595
Title: An Open Trial to Assess the Tolerability of AVANZ Olive Immunotherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-X-01; 2011-004852-20 (EudraCT Number)
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Allergic Rhinitis Due to Olea Europaea Pollen
Keywords: Olea sensitization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immunotherapy (Experimental): AVANZ
  Interventions: Biological: AVANZ olea

INTERVENTIONS:
Biological: AVANZ olea — Immunotherapy Olea europaea

SUMMARY:
This trial is an open, national, multi-centre trial. The trial will be initiated after olive pollen season 2012 and subjects will receive treatment for 6 weeks.

The aim of study is to assess the tolerability of the up-dosing phase of AVANZ Olive. The frequency of patients with adverse reactions will be the primary endpoint.

Frequency of patients with systemic reactions according to EAACI classification, increase in IgG4 and in IgE and reduction in immediate skin reactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18-65 years of age.
2. A clinical history of olive pollen induced allergic rhinoconjunctivitis with or without asthma at least one year prior to trial entry.
3. Positive SPT to olive pollen (wheal diameter ≥ 3 mm).
4. A positive specific IgE against olive pollen (≥Class 2; ≥0.70 KU/L) documented in the last 5 y

Exclusion Criteria:

1. FEV1 < 70% of predicted value at screening after adequate pharmacologic treatment.
2. Uncontrolled or severe asthma.
3. A clinically relevant history of symptomatic perennial allergic rhinitis and/or conjunctivitis caused by an allergen to which the subject is regularly exposed and sensitized.
4. History of severe asthma exacerbation or emergency room visit or admission for asthma in the previous 12 months.
5. At screening, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infection (serous otitis media is not an exclusion criterion).
6. Treatment with parenteral corticosteroids, oral corticosteroids or anti-IgE in the previous 3 months or during the study (except for steroids if needed as rescue medication).
7. Currently treated with angiotensin converting enzyme (ACE) inhibitors, tricyclic antidepressants, β-blockers, mono amine oxidase inhibitors (MAOIs) and any other drug containing alum (e.g. antacids) taken on a daily basis.
8. Previous treatment by other allergen concomitant IT or immunotherapy with Olea europaea extracts within the previous 5 years (initiation of subcutaneous immunotherapy is acceptable if treatment has been discontinued before reaching maintenance dose; for SLIT 3 months in the last 5 years is accepted).
9. History of anaphylactic shock due to e.g. food, insect venom, exercise or drug.
10. History of severe and recurrent angioedema.
11. Any contraindication according to the Investigator Brochure (IB).
12. Use of an investigational drug within 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with adverse reactions. | Participants will be followed for an expected average of 6 week.s
  From date of inclusion until date of last visit documented, it's expected an average of 6 visits, assessed up to 6 weeks per subject.

SECONDARY OUTCOMES:
Frequency of patients with systemic reactions according to EAACI classification. | Participants will be followed for an expected average of 6 weeks.
  From date of inclusion until date of last visit documented, it's expected an average of 6 visits, assessed up to 6 weeks per subject.

CONTACTS AND LOCATIONS:
Overall Officials: CARMEN MORENO, MD, Principal Investigator — HOSPITAL UNIVERSITARIO REINA SOFÍA Córdoba- Spain
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Córdoba, Spain

REFERENCES:
- [Derived] Moreno C, De San Pedro BS, Millan C, Panizo C, Martin S, Florido F. Exploratory study of tolerability and immunological effect of a short up-dosing immunotherapy phase with a standardised allergen extract derived from pollen of Olea europaea. Clin Transl Allergy. 2015 Jul 24;5:27. doi: 10.1186/s13601-015-0070-y. eCollection 2015. PMID 26213608